CLINICAL TRIAL: NCT02089711
Title: Multi-center Study for Normal Database of Optic Nerve Head, Retinal Nerve Fiber Layer, and Macula Parameters With the Heidelberg Spectralis OCT, Study 2
Brief Title: Optical Coherence Tomography (OCT) Normative Data Collection Study (S-2013-2)
Acronym: S-2013-2
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2013-2 NORM-jp
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Normal subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Japanese healthy subjects: subjects with healthy eyes

SUMMARY:
This study is being initiated to create a normal database including measures of optic nerve head (ONH), peripapillary retinal nerve fiber layer (RNFL), and macula using the Heidelberg Spectralis OCT device. The range will be determined for each structural parameter across normal eyes in Japanese subjects, and the measurements stratified according to age.

DETAILED DESCRIPTION:
This multi-center, prospective, observational (non-interventional) study is the second in a series to measure structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT device. This study is conducted in normal Japanese volunteers. The main goal of the study is to provide the range of these structural parameters in normal eyes. The study will include at least 224 (enrollment target: 249) normal volunteers; each study site will recruit 32 to 40 subjects with an age range of 18 to 90 years and an approximately equal number of females and males. All subjects will undergo Spectralis OCT imaging, biometric and ophthalmoscopic examination, disc photography and visual field testing in one single visit. All examinations performed on the subjects are non-significant risk procedures because the medical devices are cleared for marketing in Europe and in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Subject is not an employee of the eye clinic.
* Age ≥18 to 90.
* Able and willing to undergo the test procedures, give consent, and to follow instructions.
* Healthy eye without prior intraocular surgery (except cataract surgery) and without clinically significant vitreal, retinal or choroidal diseases, clinically significant diabetic retinopathy (subject may have diabetes), or disease of the optic nerve. Small Drusen are acceptable in older subjects.
* Japanese decent (self-reported).
* Negative history of glaucoma.
* Intraocular pressure ≤21mmHg.
* Best corrected visual acuity ≥0.5.
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* Axial length ≤ 26.0 mm
* Normal visual field with Glaucoma Hemifield Test and Mean Deviation within normal limits, or not abnormal visual field by judgment of the ophthalmologist.
* Clinically normal appearance of the optic disc, with normal appearing neuroretinal rim with respect to color and shape. The optic disc is examined ophthalmoscopically and by evaluation of stereo photographs.
* When both eyes are eligible, both eyes enter the study.

Exclusion Criteria:

* Unreliable visual field. The reliability indices should be used as guide as well as the perimetrist's notes.
* Unusable disc stereo photos.
* Inability to undergo the tests.
* Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance).

Minimum requirements are:

* Retina completely included in image frame,
* Quality Score ≥ 20 in the stored ART mean images, and
* For ONH-R scan: Center position error ≤ 100 μm.

Note: Inability of a subject to perform one of the two scan patterns or insufficient image quality in one scan pattern does not exclude the subject or eye from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 224 Japanese subjects (enrollment target: 249 subjects) will be selected from qualifying normal volunteers. Age ranges will be from ≥18 to 90 years. Recruitment will be from persons who respond to recruitment initiatives at the individual centers or have signed a release saying that they are willing to be approached for participation in research.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Normative data for ONH dimensions, RNFL thickness, retinal thickness and thickness of retinal layers at the macula. | 12 months
  This normal database will be used to determine if an unknown subject has measurement values "within normal limits" or "outside normal limits." It is planned to classify an eye "within normal limits" if the measurement value is greater than or equal to the 5th percentile of the normal distribution, and as "outside normal limits" if the measurement value is smaller than the 1st percentile (or larger than 99th percentile) of the normal distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Araie, MD, PhD, Principal Investigator — Tokyo University
Locations (1):
- The University of Tokyo, Tokyo, Tokyo, Japan